CLINICAL TRIAL: NCT03639350
Title: Obesity, Body Fat Distribution, and Cancer Risk in the Multiethnic Cohort Study
Brief Title: The Healthy Diet and Lifestyle Study
Acronym: HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: The William and Ellen Melohn Endowed Research Fund (Unknown)
Responsible Party: Principal Investigator, Carol J Boushey, Associate Research Professor, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12619302B; 4502286 (Other: University of Hawaii Cancer Center)
Record Dates: First submitted 2018-06-22; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Visceral Fat
Keywords: intermittent energy restriction; Randomized Controlled Trial; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Participants will be randomized to either the IER+Med diet or the DASH diet for 12 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be provided with healthful dietary information but will not be told what diets their diet plans are based on. Participants in the IER+MED diet group will be told they are on diet plan 1 and participants in the DASH diet group will be told they are on diet plan A. The research dietitians will know which diet plan each participant is on, however; all other clinic staff who assess outcomes measures will be blinded to each participant's diet group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IER+MED group (Experimental): The IER+MED group intervention will be to restrict 70% energy (34%, 33% and 33% distribution of protein, carbohydrate, and fat, respectively) on 2 days and follow the MED diet (25%, 45%, 30%) and meet their estimated energy requirement (EER) for the other 5 days each week. Participants will also be asked to follow a moderate exercise program (1 hour of walking five days a week).
  Interventions: Behavioral: IER+MED group
- DASH group (Active Comparator): The DASH group intervention will be to follow the DASH diet and meeting a distribution of macronutrients of 20% protein, 53% carbohydrate, and 30% fat and meet their EER. Participants will also be asked to follow a moderate exercise program (1 hour of walking five days a week).
  Interventions: Behavioral: DASH group

INTERVENTIONS:
Behavioral: IER+MED group — Follow a Mediterranean diet 5 days per week and follow intermittent energy restriction 2 days per week.
  Arms: IER+MED group
Behavioral: DASH group — Follow the distribution of macronutrients and food groups prescribed by the DASH diet 7 days per week.
  Arms: DASH group

SUMMARY:
This pilot study aims to develop a study design to test the difference between a fasting diet and a heart healthy diet, assess participants' adherence to the study design, and to test whether either diet helps to reduce fat wrapped around the organs in the stomach area and total body fat in East Asian American adults. 70 men and women residents of Oahu Hawai'i, aged 35-55, who are overweight or obese and have moderate to high amounts of fat around organs in the stomach area, of Japanese, Chinese, or Korean ancestry, will be equally distributed to either the fasting diet or the heart healthy diet and asked to follow this diet for the 12-week study. Each diet has set requirements for energy, protein, carbohydrates, and fat. The fasting diet has two days of fasting, where participants will be asked to follow a low carbohydrate- low energy diet, and five days of a balanced diet without any energy restriction (the Mediterranean diet). The other group will follow a heart healthy diet (Dietary Approaches to Stop Hypertension diet) for all seven days without any energy restriction. Both groups will be asked to follow a moderate exercise program (one hour of walking five days a week). Dietitians will provide information on diet and exercise requirements to the participants at the start of the study. Dietitians will contact the participants seven times, primarily by phone, to offer support and to check if the participants are following prescribed diet and exercise plans. Participants will use a mobile phone app to take images of all foods and drinks for four days at the beginning, middle and end of the 12-week study. Body measurements, including measurements of body fat, will be taken at the beginning and end of the study by trained clinic staff. The analysis of the food images, participants' self-reported compliance to diet and exercise plans, and body measurements will be used to determine if the study design and participant compliance to the study are successful, and to assess which diet is better at reducing total body fat and fat around the organs in the stomach region.

DETAILED DESCRIPTION:
Background and rationale: East Asian adults are known to have higher levels of visceral adiposity than whites, African Americans, and Hispanic adults in the US. This visceral fat deposition, because of its close proximity to the portal vein, has greater metabolic activity and is associated with a greater risk of cardiometabolic diseases and possibly certain cancers (e.g., breast and colorectal cancers). Newly introduced weight loss interventions, specifically, intermittent energy restriction (IER), have been proposed to be as effective as continuous energy restriction, achieve higher and long-term compliance, and may predominantly result in a decrease in visceral fat. Thus, implementing this novel weight loss intervention among East Asian Americans with high visceral fat deposition would be particularly beneficial .

Goal: This study aims to demonstrate the feasibility to conduct an intermittent energy restriction (IER) nutritional intervention aimed at reducing visceral adiposity in overweight Asian Americans middle-aged adults.

1. To finalize and implement a protocol for an IER intervention plus exercise with the goal of reducing visceral fat in overweight adult East Asian Americans (EAA). The protocol will include an intensive dietary intervention and an exercise program administered by a dietitian through individual meetings and the use of new technologies to monitor dietary compliance.
2. After eligibility screening, 70 individuals will be randomized to either the intensive intervention diet group or to a non-intensive intervention (active comparator) diet group for 12 weeks. The intensive intervention group will follow a low carbohydrate- low energy IER diet for two consecutive days, and the Mediterranean (MED) diet for the other five days and meet estimated energy requirements (IER + MED group). The active comparator group will follow the Dietary Approaches to Stop Hypertension (DASH) diet for all seven days and meet estimated energy requirements (DASH group). With an expected attrition rate of ~25%, the investigators expect ~50 participants to complete the study.
3. To evaluate study retention, protocol adherence, effect size of the intervention on body weight, total adiposity, DXA measured visceral fat (main outcome), estimated visceral adipose tissue area, and selected clinical measures (e.g., waist circumference, hip circumference).

Design: Randomized lifestyle intervention trial to compare the effects of two twelve-week diets - (i) an IER + MED diet versus (ii) DASH diet- on DXA quantified visceral fat deposition distribution in overweight/obese men and women. Both intervention groups will be asked to follow a moderate exercise program (1 hour of walking five days a week). The research will be carried out in the University of Hawaii Cancer Center (UHCC). The investigators will determine and compare the primary and secondary endpoints at least five days after the last 2 energy-restricted days to a corresponding day of the week in the DASH group at the completion of the 12th week of IER+MED or DASH diets.

Assessing dietary intervention adherence: Dietary intake of energy, fat (monounsaturated fatty acids (MUFA), Polyunsaturated fatty acids (PUFA) and saturated fat), carbohydrate, protein, dietary fiber and alcohol will be assessed prior to the first week of intervention, the 5-6th week, and the 12th week. Participants will capture images of foods eaten and consumed over four days (i.e., before and after images of each eating occasion). A mobile app designed to seamlessly take images of foods/beverages will be loaded to onto each participant's mobile telephones for free and removed at the end of the study. Physical activity level will be assessed at baseline using a physical activity questionnaire.

Advice, support and monitoring in both diet groups Foods eaten for the IER+MED and DASH diets will be self-selected by the participants and not provided by the study team. The IER+MED and DASH groups will receive clear instructions on how to follow the allocated diet in a face-to-face dietary consultation with one of the trial dietitians (45- 60 minute appointment) at the UHCC. Both groups will receive comprehensive written instructions of how to follow the diets at home, including recommended portion sizes and recipes and suggested meal plans. Both groups will receive appropriate behavioral techniques to promote adherence to diets (i.e., self-monitoring of diet and goal setting).

Participants will be contacted by telephone by an allocated dietitian one week after randomization to check that they have started the diet, to assess understanding of the diet and to provide any trouble shooting advice. Participants will be contacted by an allocated dietitian with weekly phone calls in weeks 1 to 4 to discuss adherence and any problems with the diet; and with every other week phone calls in weeks 5 to 12. Both groups will be asked to record 4-day dietary records with the mobile food record at Week 6 and Week 11. This will allow assessment to adherence of the allocated diets and better tailor dietary advice. Participants will be asked to report overall compliance to the diet and physical activity plans using a scale of 0-10 for each, on the weekly and fortnightly phone calls with the dietitian. The IER+MED group will also be asked to record adherence to the 2-day IER using a scale of 0-2. All participants will also be advised to become more active, walking at least one hour per day five days per week. The intermittent energy restriction (IER) group will be encouraged to walk on the non-IER days.

Post-Study At the end of the study all participants will be offered advice on continued weight loss and/or weight loss maintenance if they have reached a target weight and this is appropriate. This will include advice regarding preferred diet, i.e., IER+MED or DASH. If resources permit, the investigators will recontact participants six and twelve months after the end of the intervention to assess dietary intake, physical activity and body weight.

Statistical Considerations Statistical analysis will be conducted within Epidemiology Program, UHCC. The primary aim is to determine changes in percentage visceral fat between the IER+MED diet and the DASH diet over a 3 months period. The sample size of 25 participants per group has been chosen to detect a difference of 15 percentage points in the reduction in visceral fat between the two different diets, assuming an estimated 25% drop-out rate. Calculations assume a two-sided t-test with estimated standard deviation of 10% and the conventional 5% significance level. The primary analysis will be performed on an intent-to-treat principle, where all participants will be analyzed by randomization group, regardless of compliance.

The primary endpoints of visceral fat measurements will be regressed on randomization group and time point, as well as potential confounders, using a mixed model approach accounting for the repeated measures at baseline, and 6 and 12 weeks. The primary hypothesis will be tested by a contrast F test comparing the difference between groups in the change from baseline to 12 weeks. The 6 month assessment will be similarly tested to understand the trend over time. If there is evidence of a linear change in fat over time, time will be entered as a continuous variable and the slope will be compared between groups. Visceral fat will be modelled as an absolute area and as percentage of total area. The secondary analysis will analyze relationship between the IER+MED intervention and total adiposity.

Ethical Considerations The study will be performed in accordance with the ethical principles in the Declaration of Helsinki and the University of Hawaii operational and ethical guidelines for research and other applicable regulatory requirements.

Participant information and consent Consent to enter the study will be sought from each participant only after a full explanation has been given, information has been provided and time allowed for consideration. The right of the participant to refuse to participate without giving reasons will be respected.

Discontinuation and withdrawal Participants are free to withdraw from the study at any time, without prejudice to further treatment. Participants may also be discontinued from the study at any time, at the discretion of the investigator. Requests by the participant to be withdrawn from the study should be made through the principal investigator.

Confidentiality After the participant has consented, any information from the study will be stored on a secure password-protected computer that will be accessible only to the research team. Trial data on anthropometry and activity meter data will be kept in a secure computer at the UHCC. The food & beverage images from the 4-day mobile food records will be kept on a secure server.

Data Handling and Record Keeping All data will be kept strictly confidential. Any individual volunteering to participate will be assigned a code number, with the link to identifying information only available to the few study staff that require this information. Identifying information will be maintained in separate secure computer files from the remainder of the data. All forms will be stored in locked file cabinets, and those with identifying information will be stored separately from the other forms. No analysis will ever identify participants individually.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-40
* No serious health issues
* Normal blood chemistry profile
* VAT ≥90cm2 for men and ≥80cm2 for women
* Japanese, Chinese, or Korean ancestry
* Resident of Hawaii.

Exclusion Criteria:

* Reported smoking tobacco products or marijuana in the past 2 years
* Taking medication for Type 1 or Type 2 diabetes
* Reported taking thyroid medication.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visceral adipose tissue (VAT) at 12 weeks | Change from baseline VAT at 12 weeks
  VAT (cm2) measured at L4-L5 with Dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change from Baseline Blood Biomarkers at 12 weeks | Change from baseline blood biomarkers at 12 weeks
  Insulin, Glucose, C-reactive protein (CRP), Interleukin-6 (IL-6), Adipokines (leptin and adiponectin), Insulin-like growth factor-1 (IGF-1), and Serum Lipids
Change from Baseline DXA Subcutaneous Fat and Total Adiposity at 12 weeks | Change from baseline subcutaneous fat and total adiposity at 12 weeks
  DXA subcutaneous fat and total adiposity
Change from Baseline Lean Body Mass at 12 weeks | Change from baseline lean body mass at 12 weeks
  DXA lean body mass
Change from Baseline Resting Energy Expenditure (REE) at 12 weeks | Change from baseline REE at 12 weeks
  REE measured with indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Loic Le Marchand, MD, PhD, Principal Investigator — University of Hawaii Cancer Research Center; Carol J Boushey, PhD, RDN, Study Chair — University of Hawaii Cancer Research Center; Unhee Lim, PhD, Study Chair — University of Hawaii Cancer Research Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvie M, Wright C, Pegington M, McMullan D, Mitchell E, Martin B, Cutler RG, Evans G, Whiteside S, Maudsley S, Camandola S, Wang R, Carlson OD, Egan JM, Mattson MP, Howell A. The effect of intermittent energy and carbohydrate restriction v. daily energy restriction on weight loss and metabolic disease risk markers in overweight women. Br J Nutr. 2013 Oct;110(8):1534-47. doi: 10.1017/S0007114513000792. Epub 2013 Apr 16. PMID 23591120
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Derived] O'Reilly H, Panizza CE, Lim U, Yonemori KM, Wilkens LR, Shvetsov YB, Harvie MN, Shepherd J, Zhu FM, Le Marchand L, Boushey CJ, Cassel KD. Utility of self-rated adherence for monitoring dietary and physical activity compliance and assessment of participant feedback of the Healthy Diet and Lifestyle Study pilot. Pilot Feasibility Stud. 2021 Feb 11;7(1):48. doi: 10.1186/s40814-021-00786-3. PMID 33573693
- [Derived] Panizza CE, Lim U, Yonemori KM, Cassel KD, Wilkens LR, Harvie MN, Maskarinec G, Delp EJ, Lampe JW, Shepherd JA, Le Marchand L, Boushey CJ. Effects of Intermittent Energy Restriction Combined with a Mediterranean Diet on Reducing Visceral Adiposity: A Randomized Active Comparator Pilot Study. Nutrients. 2019 Jun 20;11(6):1386. doi: 10.3390/nu11061386. PMID 31226790